CLINICAL TRIAL: NCT00322569
Title: A Randomized, Multi-Center Study of the Pimecrolimus-Eluting (Corio™) and Pimecrolimus/Paclitaxel-Eluting Coronary Stent System (SymBio™) in Patients With De Novo Lesions of the Native Coronary Arteries
Brief Title: A Randomized, Multi-Center Study of the Pimecrolimus-Eluting and Pimecrolimus/Paclitaxel-Eluting Coronary Stent Systems (GENESIS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Collaborators: Conor Medsystems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-01
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Disease
Keywords: Percutaneous coronary intervention (PCI); Drug eluting stent (DES)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Corio™ Pimecrolimus-Eluting Cobalt Chromium Coronary Stent System
  Interventions: Device: Corio™ Pimecrolimus-Eluting Coronary Stent System
- 2 (Experimental): SymBio™ Pimecrolimus/Paclitaxel-Eluting Coronary Stent System
  Interventions: Device: SymBio™ Pimecrolimus/Paclitaxel-Eluting Coronary Stent System
- Control Arm (Active Comparator): Costar ™ Paclitaxel-Eluting Coronary Stent System
  Interventions: Device: Costar ™ Paclitaxel-Eluting Coronary Stent System

INTERVENTIONS:
Device: Corio™ Pimecrolimus-Eluting Coronary Stent System — Drug-eluting stent
  Arms: 1
Device: SymBio™ Pimecrolimus/Paclitaxel-Eluting Coronary Stent System — Drug-eluting stent
  Arms: 2
Device: Costar ™ Paclitaxel-Eluting Coronary Stent System — Drug-eluting Stent
  Arms: Control Arm

SUMMARY:
To demonstrate non-inferiority in 6-month angiographic in-stent late lumen loss of the pimecrolimus-eluting coronary stent (Corio) compared to the CoStar coronary stent control arm and the dual pimecrolimus/paclitaxel-eluting (Symbio) coronary stent compared to the CoStar coronary stent control arm for the treatment of single de novo lesions <25 mm in length in native coronary arteries 2.5 - 3.5 mm in diameter.

DETAILED DESCRIPTION:
This study is designed to evaluate 6 month in-stent late lumen loss of the 1) Corio™ pimecrolimus-eluting coronary stent system and the 2) SymBio™ dual pimecrolimus/paclitaxel-eluting coronary stent system compared to the CoStar™ Paclitaxel-Eluting Coronary Stent System control arm.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Eligible for percutaneous coronary intervention (PCI).
2. Documented stable or unstable angina pectoris
3. Left ventricular ejection fraction (LVEF) ≥25%
4. Acceptable candidate for coronary artery bypass graft surgery (CABG).
5. Target lesion < 25 mm in length with RVD of ≥2.5 mm to ≤3.5 mm with visually estimated stenosis of ≥50% and < 100% .
6. Target vessel had not undergone prior revascularization within the preceding 6 months.
7. Target lesion must have been a minimum of 10 mm distance from any previously treated segment of the target vessel
8. Patient understood the study requirements and the treatment procedures and provided written Informed Consent, approved by the local Ethics Committee.
9. Willing to comply with all specified follow-up evaluations.

Exclusion Criteria:

General Exclusion Criteria

1. Known sensitivity to pimecrolimus, paclitaxel, the polymer (PLGA) or cobalt chromium.
2. Planned treatment with any other PCI device in the target vessel(s).
3. MI within 72 hours prior to the index procedure
4. The patient is in cardiogenic shock.
5. Cerebrovascular Accident (CVA) within the past 6 months.
6. Acute or chronic renal dysfunction
7. Contraindication to ASA or to clopidogrel.
8. Thrombocytopenia
9. Active gastrointestinal (GI) bleeding within the past 3 months.
10. Any prior true anaphylactiod reaction to contrast agents
11. Patient is currently taking colchicine, chronic systemic steroid therapy or systemic immunosuppressant therapy, or or had been treated with paclitaxel (systemic) within 12 months of the index procedure.
12. Patient was currently, or was on long term intermittent therapy with topical pimecrolimus
13. Female of childbearing potential.
14. Life expectancy of less than 24 months due to other medical conditions.
15. Co-morbid condition(s)
16. Currently participating in another investigational drug or device study

General Angiographic Exclusion Criteria:

1. Left main coronary artery disease (stenosis >50%), whether protected or unprotected.
2. Target lesion was ostial in location (within 3.0 mm of vessel origin).
3. Target lesion and/or target vessel proximal to the target lesion was severely calcified by visual estimation.
4. Target lesion involved a bifurcation with a diseased (>50% stenotic) branch vessel >2.0 mm in diameter that required intervention.
5. Target lesion was totally occluded Thrombolysis In MI (TIMI flow 0) or TIMI flow ≤1.
6. Angiographic presence of probable or definite thrombus.
7. Target vessel would have been pre-treated with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon or transluminal extraction catheter immediately prior to stent placement.
8. Prior coronary intervention using brachytherapy to any segment of the target vessel.
9. The target vessel had prior drug-eluting stent placement to vessel segment (or branch) proximal to intended target lesion site within preceding 6 months.
10. Angiographic restenosis of any segment of the target vessel that had undergone prior percutaneous coronary intervention.
11. Angiographic evidence of atherosclerotic disease with >50% diameter stenosis (by visual estimate) proximal or distal to the target lesion (applies to the major epicardial portion of the target vessel and contiguous vessel segment if the target lesion was located in a branch vessel).
12. Prior surgical revascularization of the target vessel with patent graft (saphenous vein graft or arterial conduit).
13. Target lesion lied within 10mm of prior surgical anastomosis site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Primary angiographic late loss in the stent as measured by Quantitative Coronary Angiography (QCA) | 6 months post-procedure

SECONDARY OUTCOMES:
MACE (composite of non-cardiac death, new Qw/nonQw MI, and TVR) as described below | 30 days and 6 months
  Major Adverse Cardiac Events (MACE) defined as an adjudicated composite of death that cannot be clearly attributed to a non-cardiac event or non-intervention vessel, new myocardial infarction (Q-wave or non-Q-wave) that cannot be clearly attributed to a non-intervention vessel and clinically driven target vessel revascularization (TVR)
Primary Device Success defined as attainment of <50% in-stent residual stenosis of the target lesion using only the assigned device in the absence of device malfunction and device-related complication. | 30 days and 6 months, 1, 2, 3, 4, and 5 years post-procedure
Lesion Success defined as attainment of <50% residual stenosis of the target lesion using the assigned study device or any percutaneous method. | 30 days and 6 months, 1, 2, 3, 4, and 5 years post-procedure
Procedure Success defined as attainment of final lesion success in the absence of in-hospital MACE. | 30 days and 6 months, 1, 2, 3, 4, and 5 years post-procedure
Angiographic in-stent and in-segment binary restenosis (≥50% diameter stenosis). | 30 days and 6 months, 1, 2, 3, 4, and 5 years post-procedure
In-stent and in-segment MLD | 6 months post-procedure
In-segment angiographic late loss | 6 months post-procedure
Clinically driven Target Lesion Revascularization (TLR) | 6 months post-procedure
Percent volume obstruction of the stent by intravascular ultrasound (IVUS) in the IVUS cohort. | 6 months post-procedure
Incidence of late acquired incomplete stent to vessel apposition (stent malapposition) by IVUS in the IVUS cohort. | 6 months post-procedure
Incidence of reported MACE | 1, 2, 3, 4 and 5 years post-procedure
Comparison of the pimecrolimus-eluting stent to the pimecrolimus/paclitaxel-eluting stent for primary and secondary endpoints. | 30 days and 6 months, 1, 2, 3, 4, and 5 years post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Curzen, M.D., Principal Investigator — Southampton University Hospital; Stefan Verheye, M.D., Principal Investigator — AZ Middelheim Hospital
Locations (1):
- Southampton University Hospital, Southampton, United Kingdom

REFERENCES:
- [Result] Verheye S, Agostoni P, Dawkins KD, Dens J, Rutsch W, Carrie D, Schofer J, Lotan C, Dubois CL, Cohen SA, Fitzgerald PJ, Lansky AJ. The GENESIS (Randomized, Multicenter Study of the Pimecrolimus-Eluting and Pimecrolimus/Paclitaxel-Eluting Coronary Stent System in Patients with De Novo Lesions of the Native Coronary Arteries) trial. JACC Cardiovasc Interv. 2009 Mar;2(3):205-14. doi: 10.1016/j.jcin.2008.12.011. PMID 19463427